CLINICAL TRIAL: NCT00494351
Title: Prospective Controlled Study of the Efficacy of NdYag for Hidradenitis Suppurativa
Brief Title: Study on the Effect of NdYag Laser for the Treatment of Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB4309
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Nd:YAG laser
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Long-pulsed Nd:YAG laser 1064 nm — Laser once monthly
  Other Names: Long pulsed Nd:YAG laser

SUMMARY:
* Determination of the short and long term efficacy of NdYag laser for treatment of Hidradenitis suppurativa, which is an inflamed, deeper follicular disorders.
* Determination of patient tolerance of discomfort associated with NdYag laser treatment for Hidradenitis suppurativa.
* Determination of the impact of this condition on quality of life and if there is any impact of therapy in the dermatology quality of life index.
* Evaluate the histopathologic changes of YAG therapy on affected skin

Second phase of study:

* Prospective, controlled clinical and histologic study of patients with Hurley Stage II HS disease.
* 19 patients of skin types II to VI with Hurley Stage II hidradenitis suppurativa lesions of the axilla and groin. This is a different set of patients than those treated in the first phase of the study above. This study primarily focuses on and further characterizes the histologic changes after laser treatment.

DETAILED DESCRIPTION:
1. Background:

   Hidradenitis suppurativa (HS) is a chronic suppurative recurrent disease of the apocrine glands. Histological studies suggest that it is a disease of the follicles with apocrine involvement as a secondary event. There is limited efficacy of medical treatments and high morbidity for surgical treatment. Limited data are available on the short and long term efficacy of laser treatments for use in HS.
2. Purpose of the study:

   To investigate the efficacy of NdYag 1064nm laser for the treatment of hidradenitis suppurativa.
3. Significance:

   Hidradenitis suppurativa is a chronic, often suppurative skin condition which affects primarily the hair follicles. A variety of therapies have been used to treat HS, often with unsatisfactory results. As the Nd Yag laser is a highly effective laser treatment for hair removal as well as for the treatment of deeper follicular disorders of the skin which associated inflammation, we postulate that the Nd Yag may be highly effective for decreasing the inflammation, pain, suppuration and frequency of recurrence of HS.
4. Study design:

   * we are treating patients with HS Hurley Stage II on one side of the body with long-pulsed Nd:YAG laser.
   * The control is the patient's opposite symmetrical side of the body.
   * Pre-treatment assessment is performed along the Hidradenitis Suppurativa European Research Group (HISERG) scale.
   * The control will be the patient's opposite symmetrical side of the body.
   * Each patient is treated on a monthly basis for up to 4 months, and then 2 months of follow up to observe the long term effect of the treatment and to detect any relapse.
   * A study of our primary investigator on treating dissecting cellulitis, which is also a follicular disease like HS, with the long-pulsed Nd:YAG laser aimed at determination of the capabilities and limitations of this modality with respect to reducing pus formation; enabling the termination of systemic treatments; investigating the side-effect profile including dyspigmentation and scarring alopecia; and terminating the disease process. The study showed that one year after initiating laser treatment, patients achieved decreased pus formation, a reduced reliance on systemic treatments, and a controlled or terminated disease process without dyspigmentation.
5. Second phase of study:

   * Two monthly laser sessions were performed using the long-pulsed Nd:YAG 1064 nm laser on a new set of 19 patients.
   * Clinical response was scored using the modified Hidradenitis Suppurativa Lesion Area and Severity Index (LASI). Histologic changes were examined before treatment, 1 week, 1 month and 2 months post-treatment. Histologic controls were obtained from untreated, involved sites.

ELIGIBILITY:
Inclusion Criteria:

For inclusion, the subject must:

* Be at least 18 years old
* Be otherwise healthy
* Have a diagnosis of HS
* Patients with Hurley stage II, with one ore more widely separated recurrent abscesses, with a tract and scarring, bilateral and symmetrical, will be eligible for inclusion in the study.
* Agree to abide by the Investigator's guidelines regarding photosensitizing drugs
* Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
* Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

* Patients with Hidradenitis Hurley state I and III will be excluded from participation in the study.
* The control for this study will be the patient's opposite side of the body, i.e., for patients treated on the left axilla, the right axilla will serve as the corresponding control.
* Concomitant use of systemic or topical treatments for HS. Patients must discontinue all forms of oral therapy as systemic and topical antibiotics and retinoids for 2 weeks prior to the start of any treatment.
* Exacerbation of the patient's original condition expressed clinically by a shift from Hurley Stage II to Stage III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
We will be measuring patients' response by the clinical scoring criteria of the Hidradenitis Suppurativa European Research Group (HISERG) scale. | 6 months
Examining histologic changes at various time points following 1064 nm Nd:YAG laser treatment of hidradenitis suppurativa. | 6 months.

SECONDARY OUTCOMES:
Completion of a post treatment survey regarding the pain of the treatment, pain of their skin condition after treatment, frequency of breakouts, effectiveness of treatment, overall level of satisfaction, likelihood to use the treatment again. | Monthly, through 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H. Hamzavi, M.D., Principal Investigator — Department of Dermatology, Henry Ford Health System
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

REFERENCES:
- [Result] Krasner BD, Hamzavi FH, Murakawa GJ, Hamzavi IH. Dissecting cellulitis treated with the long-pulsed Nd:YAG laser. Dermatol Surg. 2006 Aug;32(8):1039-44. doi: 10.1111/j.1524-4725.2006.32227.x. PMID 16918566
- [Derived] Mahmoud BH, Tierney E, Hexsel CL, Pui J, Ozog DM, Hamzavi IH. Prospective controlled clinical and histopathologic study of hidradenitis suppurativa treated with the long-pulsed neodymium:yttrium-aluminium-garnet laser. J Am Acad Dermatol. 2010 Apr;62(4):637-45. doi: 10.1016/j.jaad.2009.07.048. PMID 20227579